CLINICAL TRIAL: NCT03639922
Title: Imatinib in Acute Ischaemic Stroke: A Phase 3, Randomized, Double-blind, Placebo Controlled, Parallel-arm Efficacy Trial of Imatinib in Acute Ischaemic Stroke
Brief Title: Imatinib in Acute Ischaemic Stroke
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Niaz Ahmed (Other)
Responsible Party: Sponsor-Investigator, Niaz Ahmed, Sponsor, Coordinating investigator, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: I-StrokeII2016; 2017-000075-85 (EudraCT Number)
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Acute Ischaemic Stroke
Keywords: acute ischaemic stroke; Imatinib; blood-brain-barrier; trombectomy; iv trombolysis
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel-arm
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study is double-blind, only after the study is completed or terminated the treatments will be made available, or if requested by the data safety board, or if requested by treating clinician in association with possible SAE/SUSAR
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imatinib (Active Comparator): Imatinib 400mg (2 tablets of 400mg) per day for 6 days
  Interventions: Drug: Imatinib 400mg
- Placebo (Placebo Comparator): 2 placebo tablets per day for 6 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Imatinib 400mg — 2 tablets of Imatinib 400mg per day for 6 days
  Arms: Imatinib
Drug: Placebo Oral Tablet — 2 tablets of placebo per day for 6 days
  Arms: Placebo

SUMMARY:
A clinical trial comparing treatment with Imatinib to placebo when administered within 8 hours of stroke onset for 6 days, in addition to conventional stroke treatment after acute ischaemic stroke.

DETAILED DESCRIPTION:
The study aims to investigate if Imatinib reduces intracerebral haemorrhage and oedema in stroke patients after IV thrombolysis and/or trombectomy. Two important complications of ischaemic stroke and its acute treatment are haemorrhage into the infarcted tissue and cerebral oedema. Leading to worsening functional outcome in survivors. Both are caused by a disruption of the blood brain barrier (BBB) by ischemia of the brain vascular endothelium and associated cells involved in maintaining the BBB. Imatinib can reduce the damage to the BBB and hence reduce the formation of oedema and haemorrhage.

The study is a phase III randomised, double-blind placebo-controlled parallel-arm trilal of patents with acute ischaemic stroke. Assessing the Clinical variables at baseline and after 3 months.

Primary objective:

To investigate if Imatinib (800 mg / day) treatment initiated within 8 hours of symptom onset and given for 6 days improves functional outcome at three months after acute ischaemic stroke

Secondary objective:

1. Investigate if Imatinib treatment improves functional outcome at three months in acute ischaemic stroke patients treated with iv thrombolysis
2. Investigate if Imatinib treatment improves neurological outcome at three months after acute ischaemic stroke
3. Investigate if Imatinib treatment improves neurological outcome at three months in acute ischaemic stroke patients treated with iv thrombolysis
4. Investigate if Imatinib reduces the frequency and grade of ICH in patients with acute ischaemic stroke treated with iv thrombolysis
5. Investigate if Imatinib reduces the frequency and grade of cerebral oedema in patients with acute ischaemic stroke treated with iv thrombolysis
6. Examine serious and non-serious adverse events in patients treated with Imatinib
7. Investigate if Imatinib reduces mortality at 3 months after acute ischaemic stroke
8. Investigate if Imatinib reduces mortality at 3 months in acute ischaemic stroke patients treated with iv thrombolysis

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of acute ischaemic stroke with a neurological deficit corresponding to 6 points or higher on the NIHSS score

   1. at the time of randomization if no recanalisation therapy performed
   2. prior to iv thrombolysis therapy alone or prior to thrombectomy alone if performed
   3. prior to iv thrombolysis if both iv thrombolysis and thrombectomy performed Ischaemic stroke is defined as an event characterised by sudden onset of acute focal neurological deficit, presumed to be caused by cerebral ischaemia and an imaging scan excluding any intracranial haemorrhage.
2. Age 18-85 years
3. Patients should be randomized as soon as possible but not later than 8 hours of symptom onset.

   1. If the patient receives iv thrombolysis alone, patient should be randomized and study drug should be given within one hour after completion of iv thrombolysis infusion
   2. If the patient receives endovascular thrombectomy (with or without prior iv thrombolysis), patient should be randomized within two hours after completion of endovascular thrombectomy and study drug given as soon as possible after randomization.
4. iv thrombolysis, if performed, is done in agreement with European Stroke Organisation guidelines and has been initiated within 4.5 hours of stroke onset (see below separate criteria for indications / contraindications)
5. Endovascular thrombectomy, if performed, is done in agreement with recently published American Stroke Association guidelines, and fulfilling the following criteria

   1. Confirmed diagnosis on Computed Tomography Angiography (CTA) or Magnetic Resonance Angiography (MRA) of acute occlusion of either of the first two segments of the Middle Cerebral Artery (M1 or M2), terminal Carotid Artery, first segment of the Anterior Cerebral Artery (A1), or Basilar Artery, consistent with the clinical symptoms.
   2. thrombectomy has been initiated within 8 hours of symptom onset (defined as start with femoral artery (groin) puncture)
6. Patient is competent to make a decision and has provided informed consent with regard to participation in the study, retrieval and storage of data and follow up procedures

Exclusion Criteria:

General

1. Imaging scans show signs of large current infarction as defined by more than 1/3 of the Middle Cerebral Artery territory or ½ of other vascular territories
2. ) Known significant pre-stroke disability (mRS ≥2)
3. Severe comorbidities such as advanced dementia (estimate pre-stroke if otherwise healthy), terminal illness, and other severe medical conditions with anticipated life expectancy less than 6 months.
4. Acute pancreatitis
5. Severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension (oesophageal varices) and active hepatitis
6. Ongoing treatment with chemotherapy
7. Drugs which may increase the plasma concentration of Imatinib - ketokonazol, itrakonazol, erythromycin and claritomycin
8. Drugs which may decrease the plasma concentration of Imatinib: Dexametason, phenytoin, karbamazepin, rifampizin, phenobarbital, fosphenytoin, primidon, Hypericum perforatum (Johannesört, St John's wort)
9. Female patients with childbearing potential, if pregnancy cannot be excluded by pregnancy test (urine point-of-care pregnancy test).
10. Patient is participating in other interventional study

Additional Exclusion criteria for patients treated with intravenous thrombolysis (IVT)

1. Severe stroke as assessed clinically by NIHSS>25
2. Administration of heparin within the previous 48 hours preceding the onset of stroke with an elevated activated thromboplastin time (aPTT) at presentation, or corresponding low-molecular heparin.
3. Patients receiving oral anticoagulants, e.g. warfarin sodium (INR>1.7) or direct oral anticoagulation: dabigatran ( aPTT>40s), apixaban, rivaroxaban.
4. Platelet count below 100,000/mm3. Significant bleeding disorder at present or within the past 6 months, known haemorrhagic diathesis.
5. History or evidence or suspicion of intracranial haemorrhage including sub-arachnoid haemorrhage
6. Systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, in spite of repeated doses of i.v. medication to reduce blood pressure below these limits.
7. History of the following conditions: prior ischemic stroke within 3 months, intra-axial neoplasm, intracranial or spinal surgery within the prior 3 months, recent severe head trauma within 3 months or unruptured intracranial aneurysm>5 mm.
8. Major surgery or significant trauma in the past 10 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Functional independency at 3 months as measured by modified Rankin Scale (mRS) Score 0-2. | 3 months post treatment
  For a positive outcome, patients in the active group treated with Imatinib 800 mg per day will have statistically significant higher functional independency compared to the control group treated with placebo.

SECONDARY OUTCOMES:
Change in mRS score at 3 months compared to baseline | At baseline and 3 months post treatment
  For a positive outcome, patients treated with Imatinib will have a favorable shift of the scale.
Frequency (%) of ICH on post-treatment imaging scan in patients undergoing IV thrombolysis and or endovascular thrombectomy. | 1 day post treatment start
Grade of ICH (COED 1-3) on post-treatment imaging scan in patients undergoing IV thrombolysis and or endovascular thrombectomy. | 1 day post treatment start
Frequency (%) of cerebral oedema on post-treatment imaging scan in patients undergoing IV thrombolysis and or endovascular thrombectomy. | 1 day post treatment start
Grade (COED 1-3) of cerebral oedema on post-treatment imaging scan in patients undergoing IV thrombolysis and or endovascular thrombectomy. | 1 day post treatment start
Serious and non-serious adverse events | 3 months post teatment
Mortality at 3 months. | 3 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Niaz Ahmed, MD PhD, Study Director — Karolinska Institutet
Locations (17):
- Sweden (17):
  - Mälarsjukhuset Eskilstuna, Eskilstuna
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Hässleholms sjukhus, Hässleholm
  - Centralsjukhuset Karlstad, Karlstad
  - Centralsjukhuset Kristianstad, Kristianstad
  - Skånes Universitetssjukhus Lund, Lund
  - Skånes Universitetssjukhus Malmö, Malmo
  - Skaraborgs sjukhus Skövde, Skövde
  - Capio S:t Görans Hospital, Stockholm
  - Södersjukhuset, Stockholm
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
  - Danderyds sjukhus, Stockholm
  - Sundsvalls Sjukhus, Sundsvall
  - Umeå University Hospital, Umeå
  - Uppsala Akademiska Sjukhus, Uppsala
  - Västmanlands sjukhus Västerås, Västerås

IPD SHARING:
Plan to Share IPD: No